CLINICAL TRIAL: NCT03099044
Title: "Effects of Two Doses of Fermented Dairy Beverage on Inflammation/Immune Function in Healthy Adults Undergoing Stressful Exercise; Compared to a Placebo Beverage"
Brief Title: "Fermented Dairy Beverage on Inflammation/Immune Function in Stressful Exercise"
Acronym: DAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dairy A Day, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 69716
Record Dates: First submitted 2017-03-15; First posted 2017-04-04 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Healthy adults; three groups: Placebo, vs Single-Dose and Double Dose of Fermented Dairy Beverage consumed for 10 days. Subjected to stressful exercise at beginning and end of study. Primary outcomes: immune/inflammatory markers. Assess changes in treatment vs placebo.
Who Masked: Investigator
Masking Description: Single blind (subjects unaware of treatment identity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Active Dose (Active Comparator): Subjects are assigned to receive a single Active beverage and a single placebo beverage.
  Interventions: Other: Single Active dose
- Double Active Dose (Active Comparator): Subjects are assigned to receive 2 doses of Active beverage.
  Interventions: Other: Double Active dose
- Placebo comparator (Placebo Comparator): Subjects are assigned to receive 2 doses of a placebo beverage.
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: Placebo comparator — Subjects consume 2 placebo beverages daily for 10 days. The dose-response controls for volume consumed.
  Arms: Placebo comparator
Other: Single Active dose — Subjects consume 1 placebo + 1 Active beverages daily for 10 days. The dose-response controls for volume consumed.
  Arms: Single Active Dose
Other: Double Active dose — Subjects consume 2 Active beverages daily for 10 days. The dose-response controls for volume consumed.
  Arms: Double Active Dose

SUMMARY:
The purpose of this pilot study is to determine the effects of a Single and Double Dose of Fermented Dairy Beverage on immune health and inflammatory status in healthy adults undergoing stressful exercise.

DETAILED DESCRIPTION:
This is a "pilot" study. A total of 45 male subjects will be randomized to receive either Active product (in 2 doses) or placebo. This is a single-blind design (subjects are unaware of product type they are receiving). Randomization is in a 1:1:1 ratio for active test product (in different doses) versus placebo. Products will consume the beverages for a 10-day period. The subjects will be subjected to a defined strenuous exercise protocol on Days 1 and 10 of the study. Blood will be collected on the exercise days (pre- and post-exercise) on Days 1 and 10.

Blood will be analyzed for markers of Immunity and Inflammation, to assess the immuno-supportive and anti-inflammatory properties of the Active product. Product acceptance and tolerability will also be assessed using a VAS scale.

Outcome analysis will be based upon changes over time (from time-point 0) for within group changes as well as between group differences. That is, study will examine differences in end-points from baseline to end-of-study; as well as differences among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males, aged 18 to 50 years of age (inclusive) at the time of screening, nonsmokers for at least 10 years at the time of screening and throughout the study.

  2. BMI between 20.0 and 34.9 kg/m2 (inclusive) at the time of screening. 3. Subject is currently exercising less than 150 minutes per week. 4. Subject is in good health and appropriate for exercise as determined by physical examination, medical history, laboratory tests, cardiac monitoring and Physical Activity Readiness Questionnaire (PAR-Q) 5. Subjects must be able to understand the study, agree to the requirements and restrictions, and be willing to give voluntary consent to participate in the study.

  6. Subject states that he is able to jog, run and/or walk on a treadmill for 60 minutes.

Exclusion Criteria:

* 1. History of any clinically significant cardiovascular (e.g., blocked coronary artery disease, hypertension, hyperlipidemia, Wolff-Parkinson-White syndrome, etc.), respiratory, endocrine (e.g., diabetes I or II, etc.), renal, hepatic, gastrointestinal, hematologic, neurologic, psychiatric, connective tissue (e.g., Marfan syndrome, etc.) disease or disorder, or any uncontrolled medical illness which in the opinion of the Investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study results.

  2. Family history of any first degree relative (mother, father, sibling, child) with myocardial infarction before age 50 or any first degree relative with sudden, unexplained cardiac death.

  3. Subject with a positive result for or history of positive test result(s) for human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen or Hepatitis C antibody.

  4. Subject has a history of cancer (except localized skin cancer without metastases) within five years prior to screening.

  5. Subject has any current orthopedic problem(s) or clinically significant history of musculoskeletal injury(ies) of the legs that the PI feels may interfere with the study exercise.

  6. Subjects who are not deemed as healthy by standard physical, medical history and other means of screen testing (vitals, blood work, etc.) per PI review and discretion.

  7. Subject who is currently taking or has taken probiotics within 30 days prior to the baseline visit.

  8. Subjects who ingests yogurt (regular, Greek or Icelandic), Kefir or any fermented dairy products four or more times per week regularly within the month prior to baseline visit.

  9. Subject who regularly consumes fermented beverages, such as Kombucha. Regular is defined as more than twice per week and for more than two-weeks consistently, within the 3 months prior to baseline visit.

  10. Subject has a known or suspected allergy or hypersensitivity to trial product(s), including lactose intolerance and or dairy allergies or related product(s).

  11. Subject exhibits evidence of hepatic or renal dysfunction as evidenced by ALT or AST being ≥ 2 times the upper limit of normal or serum creatinine value ≥ 2.0 mg/dl or other clinically significant abnormal clinical laboratory value per PI discretion.

  12. Abnormal electrocardiogram (ECG) results thought to be potentially clinically significant according to the Investigator, or QT prolongation, as evidenced by QTcF >450 msec.

  13. Subject has a recent history (within 12 months of Screening) of substance or alcohol abuse.

  14. Subject has taken an investigational product within 30 days of study enrollment (Visit 1).

  15. Subject who is currently taking any concomitant medications, including prescription or over the counter (OTC), herbal or dietary supplements, vitamin and/or mineral supplements, or NSAIDS or any other anti-inflammatory products, from 7 days prior to baseline and throughout the study (other than study products).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Changes in Inflammatory and immune biomarkers o IL-6, IL-10, IL-1 beta and TNF-alpha | Days 1 and 10 of study
  IL-6, IL-10, IL-1 beta and TNF-alpha; IgA, IgG, IgM, absolute neutrophil count, absolute lymphocytes, absolute monocytes, and other immune cells.
  As there are multiple variables, statistical Outcome analysis for "within and between group differences" will be based upon changes over time (from time-point 0) for within group changes [in each outcome measure] as well as between group differences. P value for significance is set at P< 0.05 for significance and will include 95% Confidence Intervals where appropriate. As this is a pilot study, no corrective factors for multiple sets of analysis will be employed.

SECONDARY OUTCOMES:
Ease of consumption (tolerability) of products | Day 10 of study
  Product ease of consumption (tolerability) will be measured by a Visual Analog Scale. On the VAS scale of 1-10, each subject is asked: "How would you rate your tolerability, your acceptance of this product?" This will be done to compare tolerability of the two product types.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Smith, M.D., Principal Investigator — QPS Bio-Kinetic Clinical Applications, LLC
Locations (1):
- QPS Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no such plan.